CLINICAL TRIAL: NCT07273968
Title: Clinical Study Evaluating the Effect of Virtual Reality on Reducing Anxiety in Patients Undergoing Wisdom Teeth Extraction
Brief Title: Clinical Study Evaluating the Effect of Virtual Reality on Reducing Patients' Anxiety During Wisdom Teeth Extraction
Acronym: SEREIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9832
Record Dates: First submitted 2025-11-25; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Dental Anxiety; Third Molar Extraction; Oral Surgery
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Wisdom tooth extraction under local anesthesia with immersive VR hypnosis (HypnoVR® system).
  Interventions: Device: Virtual reality HypnoVR® (VR headset + hypnotic software)
- Control Group (No VR) (Active Comparator): Wisdom tooth extraction under local anesthesia alone (no VR).
  Interventions: Other: Control Group (No VR)

INTERVENTIONS:
Device: Virtual reality HypnoVR® (VR headset + hypnotic software) — CE-marked class I device combining VR immersion with hypnotic text and music therapy to reduce anxiety and pain during oral surgery.
  Arms: Virtual Reality Group
Other: Control Group (No VR) — local anesthesia alone (no VR)
  Arms: Control Group (No VR)

SUMMARY:
Dental anxiety is common during third molar extractions and may exacerbate pain perception. Local anesthesia does not prevent exposure to stress-inducing stimuli. Virtual reality (VR) combined with hypnotic scripts (HypnoVR®) provides immersive multisensory distraction. This study tests whether VR reduces perioperative anxiety and postoperative pain compared to local anesthesia alone.

ELIGIBILITY:
Inclusion criteria:

* Age 18-65
* Indication for extraction of 4 wisdom teeth or ≥2 mandibular wisdom teeth
* ASA I-II
* Written informed consent.

Exclusion criteria:

* Visual/hearing impairment
* Psychiatric disorders or psychotropics (<8 weeks)
* Claustrophobia
* Heavy smoking >10 cig/day
* Previous radiotherapy (jaw)
* ASA III-IV
* Pregnancy
* Antithrombotic therapy
* Chemotherapy
* Bisphosphonates
* Uncontrolled diabetes
* Severe anxiety requiring GA or pharmacological sedation
* No health insurance affiliation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety reduction (MDAS questionnaire) | Day 1
  5-item validated scale, score range 5-25
Anxiety reduction (MDAS questionnaire) | Month1
  5-item validated scale, score range 5-25

IPD SHARING:
Plan to Share IPD: No